CLINICAL TRIAL: NCT07014865
Title: Factors Associated With Health-related Quality of Life and Social Participation of Patients With Multiple Myeloma and Their Caregivers: a Mixed Methods Study
Brief Title: Factors Associated With Health-related Quality of Life and Social Participation of Patients With Multiple Myeloma and Their Caregivers
Acronym: MMYLIFE
Status: Recruiting | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: 121/2025/OSS/AUSLRE
Record Dates: First submitted 2025-05-20; First posted 2025-06-11 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-06

CONDITIONS: Multiple Myeloma (MM); Hematologic Neoplasm
Keywords: Quality of Life; Social Participation; Caregivers; Observational study; Qualitative Research
MeSH Terms: conditions — Multiple Myeloma; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with Multiple Myeloma: This cohort includes individuals diagnosed with multiple myeloma and receiving treatment at the Hematology Unit of the Azienda USL-IRCCS di Reggio Emilia. The cohort will reflect a real-world clinical population, including individuals across different treatment lines and sociodemographic backgrounds. Patients with severe cognitive or psychiatric comorbidities that prevent active participation (e.g., dementia, severe mental illness) will be excluded.
- Informal Caregivers of Individuals with Multiple Myeloma: This cohort will include informal (unpaid) primary caregivers of individuals with multiple myeloma who are participating in the study. For each eligible patient, we will ask if there is a caregiver-identified by the patient-available and willing to participate. Informal caregivers may include family members, relatives, or close companions who provide regular, unpaid care and support. If no caregiver is available or willing to participate, the patient may still take part in the study; however, caregivers cannot be enrolled independently of the patient.

SUMMARY:
Individuals with multiple myeloma (MM) are vulnerable because of the effects of systemic organ damage and the side effects of treatment. A decline in patients' health-related quality of life (HRQoL) and a compromised participation in everyday life was reported. The diagnosis of MM negatively affects the principal informal caregiver. This is a concurrent exploratory mixed methods study that involves the use of a quantitative and a qualitative approach. For the quantitative study, aims are to describe any possible relation between the identified factors with HRQoL and participation in individuals with MM and with reactions to caring and self-efficacy of caregivers. For the qualitative study, aims are to investigate "how" and "why" the disease impacts the daily life of individuals with MM and their caregivers. The final analyses will be based on the comparison of the results of the quantitative phase and the results of the qualitative phase.

DETAILED DESCRIPTION:
MM is a hematological disease caused by an uncontrolled proliferation of plasma cells. Individuals with MM are vulnerable because of the effects of systemic organ damage and the side effects of treatment. A decline in patients' functional status, the deterioration of health-related quality of life (HRQoL) and a compromised participation in everyday life was reported. Moreover, the diagnosis of MM occurs within the context of a family and it negatively affects the principal informal caregiver.

According to the International Classification of Functioning, Disability and Health, participation in daily life plays a key role in rehabilitation as it confers a sense of normalcy to life. Comprehensive rehabilitation intervention aiming at improving HRQoL and facilitating participation has never been implemented with this aim.

From previous systematic reviews, it emerges that patient reported outcomes (PRO) of individuals with MM have been studied mainly in randomized clinical trials, but also few observational studies have been published, conducting also in Italy. In the province of Reggio Emilia, population-based data concerning the HRQoL of individuals with MM have never been collected, as well as for their caregivers. Needs related to participation in everyday life of individuals with MM and their caregivers were mainly studied through qualitative approach.

Although qualitative data are essential in describing a phenomenon, it is currently not possible to quantify the degree of loss of participation in everyday life or to identify patients most at risk of social isolation. As a counterpart, qualitative approach may explain those situations that quantitative approach cannot verify (e.g., reasons behind conditions of social vulnerability). For these reasons, it seems appropriate to explore the patients' perceived HRQoL and participation from both quantitative and qualitative perspectives, as well as the caregivers' burden, by integrating these data. In this study, needs and difficulties in accomplishing the relevant activities and roles as well as the description of factors that act as facilitators or barriers to HRQoL and participation will be identified to screen patients that might benefit most from rehabilitation. Based on these data, comprehensive and tailored rehabilitation may be planned in future studies and tested for its impact on HRQoL and participation.

This is a concurrent exploratory mixed methods study that involves the use of a quantitative and a qualitative approach. The quantitative is the main study, while the qualitative is the sub-study. Participants of the qualitative study will be a sub-group of those recruited in the quantitative study. In this mixed methods study, we will recruit individuals with MM and caregivers.

For the quantitative study, aims are to describe any possible relation between the identified factors with HRQoL and participation in individuals with MM and with reactions to caring and self-efficacy of caregivers. Data collection will be performed through an individual semi-structured interview conducted in person, remotely or through self-administration, based on participant preference and availability.

As for individuals with MM, the semi-structured interview will consist in the collection of sociodemographic and work-related characteristics, while the side effects of treatments, the needs perceived from this population and the outcomes of interest will be collected through validated assessment tools. Disease-related factors will be retrieved from medical records.

As for caregivers, the semi-structured interview will consist in the collection of sociodemographic and work-related characteristics, while the outcomes of interest will be collected through validated assessment tools. The analyses of the quantitative phase will be carried out at the end of the quantitative data collection.

Qualitative Sub-Study To complement the findings of the primary quantitative study, a qualitative sub-study will be conducted to deepen the understanding of the disease-related experiences of individuals with MM and their informal caregivers and its consequences on daily life.

This qualitative sub-study is embedded within the larger concurrent exploratory mixed methods design. Participants in the qualitative phase will be a purposeful sub-sample of those already enrolled in the quantitative study, selected to ensure variation in the line of therapy (LOT), gender, and occupational status. Inclusion will aim to represent diverse patient and caregiver experiences.

In this qualitative sub-study, open-ended questions will be asked to participants by using interview guides, one for individual with MM and one for caregiver. Before conducting the qualitative interviews, a preliminary phase will be organized where researchers will involve expert patients and caregivers to support them in defining themes and questions of the interview guide. As an example, questions of the final interview guide will be: "Could you describe your life experience and your health after being diagnosed with multiple myeloma? How do the symptoms and the disease affect your daily life? What does caring for your loved one mean to you?".

Data will be collected through semi-structured interviews conducted in person or via video call, based on participant preference and availability. All interviews will be audio-recorded, transcribed verbatim, and analyzed through the reflexive thematic analysis using an inductive approach associated to open coding. Analysis will be iterative and involve multiple researchers to ensure inter-rater reliability of the coding procedure and the methodological rigor of the analysis.

The qualitative phase analyses will be carried out at the end of each interview because, based on the themes that will emerge from each interview, we will understand when to stop recruiting.

The final analyses of the mixed methods study will be based on the comparison of the results of the quantitative phase and the results of the qualitative phase. The comparison will be performed using data triangulation or other methods depending on the level of agreement of results of both phases. From the comparison we would like to understand to what extent the results of the qualitative study confirm those of the quantitative study or if the themes that we will develop from the qualitative interviews will show other issues. This merging of the results will allow us to define a set of criteria to identify those individuals with MM and caregivers in need of support and who could benefit more from a tailored rehabilitation intervention.

ELIGIBILITY:
Inclusion criteria for individuals with MM will be:

1. diagnosis of MM
2. adulthood (≥ 18 years)
3. in treatment (LOT I, II, or ≥ III) at the Hematology Unit
4. speak Italian fluently

Exclusion Criteria:

Comorbidities that limit collaboration (e.g., dementia, severe psychiatric disorders).

_________________________________________________________________

Inclusion criteria for caregiver will be:

1. having a loved one (individual with MM) who have participated in the quantitative phase
2. being the primary informal caregiver
3. adulthood (≥ 18 years)
4. speak Italian fluently

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult individuals diagnosed with MM who are receiving treatment at the Hematology Unit of the Azienda USL-IRCCS of Reggio Emilia, and their primary informal caregivers. This population reflects a real-world clinical context, including patients at different lines of therapy (LOT I, II, or ≥III) and with diverse sociodemographic and clinical backgrounds.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life (HRQoL) | 24 months
  HRQoL in individuals with MM measured by the European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 (Quality of Life Questionnaire - Core 30).
  The QLQ-C30 is composed of three subscales: global health status (two items), functional scales (15 items), symptom scale/ individual items (13 items). Each item is assigned a score between 1 and 4 (4-point Likert scale), excluding items n. 29 and n. 30 (7-point Likert scale). All the subscales and single-item measures range in score from 0 to 100. The higher the score for the global health status, the better the quality of life. The higher the score for the functional scale, the higher the level of functioning. Instead, the higher the score for symptom scale/items, the worse the symptoms.
Health related quality of life (HRQoL) | 24 months
  HRQoL in individuals with MM measured by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Multiple Myeloma Module (EORTC) QLQ-MY20.
  The QLQ-MY20 consists of two subscales on disease symptoms (6 items) and side-effect of treatment (10 items), one functional scale on future perspective (3 items), and one single item on body image. All the subscales and single-item measures of the QLQ-MY20 range in score from 0 to 100. A higher score for disease symptoms and side-effects of treatment indicated worse outcomes, while a higher score in the body image and future perspective indicated better outcomes.
Participation | 24 months
  Participation in individuals with MM measured by the World Health Organization Disability Assessment Schedule (WHODAS 2.0). WHODAS 2.0 captures the level of functioning in six domains of life: cognition (6 items), mobility (5 items), self-care (4 items), getting along (5 items), life activities (8 items), participation (8 items). Each item of the WHODAS 2.0 is assigned a score between 1 and 5 (5-point Likert scale). The higher the score, the higher the level of disability.
Reactions to caring | 24 months
  Reactions to caring in caregivers of individuals with MM measured by the Caregiver Reaction Assessment scale (CRA). The CRA is composed of 24 items categorized in 5 subscales: impact on schedule (5 items), impact on finances (3 items), lack of family support (5 items), impact on health (4 items) and caregiver esteem (7 items). Each item is assigned a score between 1 and 5 (5-point Likert scale). The higher the score for the impact on schedule, impact on finances, lack of family support, and impact on health domains, the more the negative impact of caregiving activity, while a higher score in the caregiver esteem domain indicated more positive impact of caregiving activity.
5. Self-efficacy | 24 months
  Self-efficacy in caregivers of individuals with MM measured by the Caregiver Inventory (CGI-I). It is composed of 21 items categorized in four subscales: managing medical information (3 items), caring for the care recipient (7 items), caring for oneself (5 items), managing difficult interactions/emotions (6 items). Each item is assigned a score between 1 and 9 (9-point Likert scale). Higher scores indicate greater self-efficacy for caregiving.
Open-ended questions of a semi-structured interview that was written by researchers and clinicians and with the support of expert individuals with MM and their caregivers to collect the disease-related experiences and its consequences on daily life | 24 months
  Themes describing the disease-related experiences and its consequences on daily life of individuals with MM and their caregivers generated through the listening of their narratives

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Unità Sanitaria Locale Reggio Emilia - IRCCS, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bates-Fraser LC, Mills J, Mihas P, Wildes TM, Kent EE, Erisnor G, Adams L, Grant SJ. "A lot to manage and still have some kind of a life": How multiple myeloma impacts the function and quality-of-life of Black-White patient-caregiver dyads. J Am Geriatr Soc. 2023 Oct;71(10):3208-3220. doi: 10.1111/jgs.18482. Epub 2023 Jun 16. PMID 37326501
- [Background] Federici S, Meloni F, Mancini A, Lauriola M, Olivetti Belardinelli M. World Health Organisation Disability Assessment Schedule II: contribution to the Italian validation. Disabil Rehabil. 2009;31(7):553-64. doi: 10.1080/09638280802240498. PMID 19191060
- [Background] Efficace F, Gaidano G, Petrucci MT, Niscola P, Cottone F, Codeluppi K, Antonioli E, Tafuri A, Larocca A, Potenza L, Fozza C, Pastore D, Rigolin GM, Offidani M, Romano A, Kyriakou C, Cascavilla N, Gozzetti A, Derudas D, Vignetti M, Cavo M. Association of IMWG frailty score with health-related quality of life profile of patients with relapsed refractory multiple myeloma in Italy and the UK: a GIMEMA, multicentre, cross-sectional study. Lancet Healthy Longev. 2022 Sep;3(9):e628-e635. doi: 10.1016/S2666-7568(22)00172-6. PMID 36102777
- [Background] LeBlanc MR, Bryant AL, LeBlanc TW, Yang Q, Sellars E, Chase CC, Smith SK. A cross-sectional observational study of health-related quality of life in adults with multiple myeloma. Support Care Cancer. 2022 Jun;30(6):5239-5248. doi: 10.1007/s00520-022-06943-5. Epub 2022 Mar 9. PMID 35262791
- [Background] Levasseur M, Lussier-Therrien M, Biron ML, Raymond E, Castonguay J, Naud D, Fortier M, Sevigny A, Houde S, Tremblay L. Scoping study of definitions of social participation: update and co-construction of an interdisciplinary consensual definition. Age Ageing. 2022 Feb 2;51(2):afab215. doi: 10.1093/ageing/afab215. PMID 35134843
- [Background] Pritlove C, Jassi M, Burns B, McCurdy A. The work of managing multiple myeloma and its implications for treatment-related decision making: a qualitative study of patient and caregiver experiences. BMC Cancer. 2021 Jul 8;21(1):793. doi: 10.1186/s12885-021-08527-8. PMID 34238260